CLINICAL TRIAL: NCT05489172
Title: Mobile Health App to Reduce Diabetes in Latina Women With Prior Gestational Diabetes
Brief Title: Mobile Health App to Reduce Diabetes in Latina Women With Prior Gestational Diabetes II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R44MD009454B; R44MD009454 (NIH)
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-07

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Single arm study to evaluate the effectiveness of Hola Bebe application (Other): Participants will receive the handout "It's never too early to prevent diabetes" and will meet with the health educator at their CHC and download the Hola Bebe app. The health educator will advise participants to watch one module and complete an action plan for each of the first 12 weeks of study and encourage participants to weigh themselves weekly. The app includes the following features:1) educational/ behavioral audio visual modules, with automatic prompting to complete an action plan at the end of each module; 2) a motivational message library so that participants can chose which motivational texts they wish to receive, how often and time of day; 3) a community forum where participants can interact with each other and ask questions to the health educator; 4) tracking of weights to allow participants to see a graphic of their weight over time by inputting weekly weights; and 5) awards program where participants can earn badges for completing modules.
  Interventions: Behavioral: Hola Bebe

INTERVENTIONS:
Behavioral: Hola Bebe — Participants will receive the handout "It's never too early to prevent diabetes" and will meet with the health educator at their CHC and download the Hola Bebe app. The health educator will advise participants to watch one module and complete an action plan for each of the first 12 weeks of study and encourage participants to weigh themselves weekly. The app includes the following features:1) educational/ behavioral audio visual modules, with automatic prompting to complete an action plan at the end of each module; 2) a motivational message library so that participants can chose which motivational texts they wish to receive, how often and time of day; 3) a community forum where participants can interact with each other and ask questions to the health educator; 4) tracking of weights to allow participants to see a graphic of their weight over time by inputting weekly weights; and 5) awards program where participants can earn badges for completing modules.

SUMMARY:
The investigators will conduct a pre-post study to evaluate the effectiveness of the Hola Bebe intervention on improving self-efficacy for healthy eating and physical activity, and on weight loss among Hispanic women with recent GDM. The Hola Bebe app provides a unique opportunity to provide an effective, culturally tailored lifestyle modification program. The investigators will provide training to health educators at the two participating sites to ensure consistency and fidelity of implementation.

DETAILED DESCRIPTION:
The study builds on the investigators' previous research in which the investigator developed a culturally-tailored Spanish and English app for Latinas with recent GDM based on Social Cognitive Theory and Behavioral Economics.

The app-based program included 12 audio/visual behavioral and educational modules on healthy eating and physical activity, motivational texts, weight tracking, personalized action plans, tiered badges, videos (easy at-home exercises, user-friendly, easy-to-follow recipes, and building a balanced plate), and an online community to communicate with other participants. All content was in plain-language Spanish and English, with Spanish and English audio voice-over. Graphics were dynamic and incorporated culturally sensitive.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Self-identify as Latina;
* Overweight or obese (BMI > or =25);
* Age 18 to 45;
* Having had a pregnancy complicated by GDM within the prior 5 years.

Exclusion Criteria:

* Currently has a diagnosis for diabetes (type 1, type 2 or secondary form);
* Has underlying disease or treatment that might interfere with participation in or completion of the protocol (e.g., cancer, moderate or severe cardiovascular disease, HIV positive, active tuberculosis, lung disease, significant gastrointestinal conditions, renal disease, major psychiatric disorders, and other at the discretion of the study clinician);
* Has diseases associated with glucose metabolism;
* Takes certain medications (e.g., glucocorticoids) which interfere with glucose metabolism.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Sallis Self Efficacy for Healthy Eating | up to 6 months
  The investigators will use the eat habits confidence survey, which includes a list of things people might do while trying to change their eating habits. The investigators are mainly interested in salt and fat intake. There are 20 items to be scored in this survey. Exapmle questions are: 1. Stick to your low fat, low salt foods when you feel depressed, bored, or tense; 2. Stick to your low fat, low salt foods when there is high fat, high salt food readily available at a party.
  The four factors for the Self-Efficacy and Eating Habits Survey should be scored as follows:
  Sticking to it: mean items I - 5 Reducing calories: mean items 6 - 10 Reducing salt: mean items 11 - 15 Reducing fat: mean items 16 - 20
Sallis Self Efficacy for Physical Activity | up to 6 month
  The investigators will use the exercise confidence survey, which includes list of things people might do while trying to increase or continue regular exercise. The investigators are interested in exercises like running, swimming, brisk walking, bicycle riding, or aerobics classes.
  There are 12 items to be scored in this survey (continued from the 1st eating habit survey).
  Example questions are: 1. Get up early, even on weekends, to exercise; 2. Stick to your exercise program after a long, tiring day at work; 3. Exercise even though you are feeling depressed.
  24. Set aside time for a physical activity program; that is, walking, jogging. swimming, biking, or other continuous activities for at least 30
  The two factors for the Self-Efficacy and Exercise Habits Survey should be scored as follows:
  Sticking to it: mean items 22, 23, 25, 26, 28 - 31 Making time for exercise: mean items 21, 24, 27, 32

SECONDARY OUTCOMES:
Weight loss | up to 6 months
  The secondary outcome compares differences between T1 and T2 for percentage of baseline weight loss, calculated by subtracting weight at end of study dividing by baseline weight.

OTHER OUTCOMES:
HbA1C level | up to 6 months
  The exploratory outcome compares differences between T1 and T2 for HbA1C levels.

CONTACTS AND LOCATIONS:
Overall Officials: Dharma Cortes, Principal Investigator — Environment and Health Group, Inc.
Locations (3):
- United States (3):
  - Environment and Health Group, Cambridge, Massachusetts
  - Brookside Community Health Center, Jamaica Plain, Massachusetts
  - Lynn Community Health Center, Lynn, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided